CLINICAL TRIAL: NCT02216838
Title: Treatment of Facial Flushing With Botulinum Toxin A Injections: A Split-Face, Double-blinded, Randomized Control Trial
Brief Title: Treatment of Facial Flushing With Botulinum Toxin A Injections
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU97514
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Facial Flushing
MeSH Terms: conditions — Blushing | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- botulinum toxin A (Experimental): This study is randomized, which means the subject will be randomly assigned (like a flip of a coin) to receive botox on the right or left side of the face and saline injections on the other side. Only one side of the face will receive botox injections.
  Interventions: Drug: botulinum toxin A
- Saline Control (Placebo Comparator): This study is randomized, which means the subject will be randomly assigned (like a flip of a coin) to receive botox on the right or left side of the face and saline injections on the other side. Only one side of the face will receive botox injections.
  Interventions: Other: Saline Control

INTERVENTIONS:
Drug: botulinum toxin A — A total of 10U will be injected at 1cm increments by the blinded dermatologist into the respective randomized side.
  Other Names: Botox
  Arms: botulinum toxin A
Other: Saline Control — A total of 0.5cc benzyl alcohol containing saline will be injected at 1cm increments by the blinded dermatologist into the respective randomized side
  Arms: Saline Control

SUMMARY:
The purpose of this study is to find out if botulinum toxin A (botox®) can be used to treat facial flushing.

This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-65 years of age with persistent facial flushing
2. Willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the study staff.

Exclusion Criteria:

1. Unable to understand the protocol or give informed consent
2. Younger than 18 or older than 65 years of age
3. Females who are pregnant or lactating
4. Known hypersensitivity to BTX-A
5. Subjects using medications that interfere with neuromuscular functions (such as aminoglycoside antibiotics)
6. Subjects who have a history of congestive heart failure, carcinoid syndrome, mastocystosis, or renal cell carcinoma
7. Botulinum toxin injections in the past 6 months
8. Ablative laser procedure in the past 6 months
9. Radiofrequency device treatment in the past 6 months
10. Ultrasound device treatment in the past 6 months
11. Medium to deep chemical peel in the past 6 months
12. Temporary soft tissue augmentation material in the area to be treated in the past year
13. Semi-permanent soft tissue augmentation material in the area to be treated in the past 2 years
14. Permanent soft tissue augmentation material in the area to be treated
15. Is planning to receive within the next 6 months, any cosmetic procedure (such as any chemical peels, botulinum toxin injections, ablative or non-ablative laser procedures, filler injections, radiofrequency procedures, dermabrasion, ultrasound and face lifting procedures) in the forehead or glabellar region.
16. Is planning to use tretinoin or retinoic acid in the next 6 months
17. Has an active infection in the forehead or glabellar region (excluding mild acne)
18. Is allergic to cow's milk protein
19. Is allergic to albumin
20. Is currently using anticoagulation therapy
21. Has a history of bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Spectrophotometer measurement | Baseline and 8 weeks
  Spectrophotometer measurement as the percent resolution on each follow up visit compared to baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States